CLINICAL TRIAL: NCT04223310
Title: Clinical Usefulness of Virtual Antiarrhythmic Drug Test in Patients With Recurred AF After Catheter Ablation(CUVIA-AF3)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-1049
Record Dates: First submitted 2019-12-20; First posted 2020-01-10 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
Keywords: Recurred Atrial Fibrillation After AFCA; AF catheter ablation; Virtual antiarrhythmic drug test
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual AAD TEST group (Experimental): 1. Perform virtual AAD test using a voltage map acquired during de novo AF ablation procedure
  2. Preselect drug with optimal antiarrhythmic effects in the patient.
  3. Take an AAD selected by virtual AAD simulation in patients who recur AF after catheter resection
  4. Drug selection should be decided according to the guidelines.
  5. A follow-up of rhythm follow-up has to be conducted according to the above study design.
  Interventions: Drug: Virtual AAD TEST group
- Empirical AAD group (Active Comparator): 1. Perform virtual AAD test using a voltage map acquired during de novo AF ablation procedure
  2. Selection of AAD based on the experience of the attending physician, independent of the results of the virtual AAD test in patients who recur AF after catheter resection
  3. Drug selection should be decided according to the guidelines.
  4. A follow-up of rhythm follow-up has to be conducted according to the above study design.
  Interventions: Drug: Empirical AAD group

INTERVENTIONS:
Drug: Virtual AAD TEST group — 1. Perform virtual AAD test using a voltage map acquired during de novo AF ablation procedure
  2. Preselect drug with optimal antiarrhythmic effects in the patient.
  3. Take an AAD selected by virtual AAD simulation in patients who recur AF after catheter resection
  4. Drug selection should be decided according to the guidelines.
  5. A follow-up of rhythm follow-up has to be conducted according to the above study design.
  Arms: Virtual AAD TEST group
Drug: Empirical AAD group — 1. Perform virtual AAD test using a voltage map acquired during de novo AF ablation procedure
  2. Selection of AAD based on the experience of the attending physician, independent of the results of the virtual AAD test in patients who recur AF after catheter resection
  3. Drug selection should be decided according to the guidelines.
  4. A follow-up of rhythm follow-up has to be conducted according to the above study design.
  Arms: Empirical AAD group

SUMMARY:
Catheter ablation for atrial fibrillation (AF) is an effective rhythm control method that shows superior rhythm outcome than antiarrhythmic drug (AAD) treatment in drug-resistant AF. However, AF catheter ablation still has a substantial recurrence rate.

The current AAD use guidelines for AF management focus on the safety of drug use. However, if the AAD efficacy evaluation system using computer modeling reflecting the individual anatomy, electrophysiology, and histological characteristics of patients is practical, it will help to select a more effective AAD type or dose.

The purpose of this study is to conduct a prospective randomized clinical study on the efficacy and safety of computer modeling for optimal AAD selection in patients with recurrent AF after catheter ablation. The investigator will evaluate the efficacy of AAD simulations by comparing virtual AAD effect guided therapy and empirical AAD use in patients with recurrent AF after AF catheterization.

The investigator will test the virtual AAD effects in the computer simulations integrated by cardiac images and 3D electrophysiological maps obtained during de novo AF ablation. The investigator will compare the effects of the most potent AAD selected by virtual AAD simulation with those of empirical AAD.

DETAILED DESCRIPTION:
A. Study design

1. Prospective randomization (Virtual AAD TEST group vs. Empirical AAD group )
2. Target number of subjects: 300 (150 per group)
3. Rhythm FU : 2012 ACC/AHA/ESC guidelines (Holter monitoring at the baseline, 2 month, and thereafter every 6 months; ECG if the patient has any symptom)
4. Anticoagulant therapy followed by 2014 ACC/AHA/ESC guidelines
5. All complications in each group will be evaluated including the re-hospitalization rate, cardioversion frequency, major cardiovascular event, and mortality rate.

B. Progress and rhythm/ECG follow-up

1. To be performed in accordance with the 2012 ACC/AHA/HRS guidelines for AF management
2. Follow-up at 2 weeks, 2 months, and thereafter every 6-month after medication.
3. Rhythm control at 2 months, and thereafter every 6-month follow-up with Holter after medication
4. If the patient complains of symptoms, ECG will be performed at any time, and rhythm follow-up will be carried out with a Holter or event recorder.

C. Follow-up All the patients will be followed-up at 2 weeks, 2, 6 months, and thereafter every 6 months. If the patient shows any symptom within the clinical study period, patient will visit the outpatient clinic. ECG will be performed at every outpatient visits, and 24-hour Holter or event recording will be performed 2months and every 6 months for 2 years, and every year after 2 years (2012 Heart Rhythm Society/EHRA/European Cardiac Arrhythmia Society Expert Consensus Statement guidelines). If atrial fibrillation or atrial tachycardia lasting more than 30 seconds is observed in 12-lead ECG or Holter, it will be evaluated as recurrence. Recurrence within 3 months after the procedure will be classified as early recurrence, and that after 3 months will be classified as clinical recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with 20~80 years old those recurred AF after catheter ablation
2. Patients who are suitable for sinus rhythm conversion and maintenance using AAD medications
3. Patients who had no history of serious side effects due to AAD medications before the procedure

Exclusion Criteria:

1. Permanent AF Patients
2. AF associated with significant structural heart disease with severe anomaly or hemodynamic effects
3. Patients expected to have serious side effects when using AAD due to sinus node dysfunction
4. Severe liver or renal failure
5. Patients with past cardiac surgery history
6. Patients who are unable to oral medication or have electrolyte abnormalities
7. Patients with active internal bleeding
8. Contraindications for anticoagulant therapy (administered anticoagulant drugs to prevent cerebral infarction) or AAD
9. Valvular AF (mitral stenosis> grade 2, mechanical valve, mitral valve repair)
10. Severe concomitant illness
11. Patients expected to live for less than one year
12. Patients with drug or alcoholism
13. Those who cannot read the agreement (literacy, foreigners, etc.)
14. Patients judged to be inappropriate for participation in clinical trials by other researchers' judgment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluation: clinical recurrence rate | At 2 months after medication
  Defined as atrial fibrillation or atrial tachycardia > 30 sec after medication within 2 year. Based on the 2012 ACC/AHA/HRS guidelines, 24-hour Holter ECG monitoring will be performed at 2 month and every 6 months, and ECG and monitoring with a Holter or an event recorder will be performed at any time if the patient complains of symptoms
Efficacy evaluation: clinical recurrence rate | At 6months after medication
  Defined as atrial fibrillation or atrial tachycardia > 30 sec after medication within 2 year. Based on the 2012 ACC/AHA/HRS guidelines, 24-hour Holter ECG monitoring will be performed at 2 month and every 6 months, and ECG and monitoring with a Holter or an event recorder will be performed at any time if the patient complains of symptoms
Efficacy evaluation: clinical recurrence rate | At 12 months after medication
  Defined as atrial fibrillation or atrial tachycardia > 30 sec after medication within 2 year. Based on the 2012 ACC/AHA/HRS guidelines, 24-hour Holter ECG monitoring will be performed at 2 month and every 6 months, and ECG and monitoring with a Holter or an event recorder will be performed at any time if the patient complains of symptoms
Efficacy evaluation: clinical recurrence rate | At 18 months after medication
  Defined as atrial fibrillation or atrial tachycardia > 30 sec after medication within 2 year. Based on the 2012 ACC/AHA/HRS guidelines, 24-hour Holter ECG monitoring will be performed at 2 month and every 6 months, and ECG and monitoring with a Holter or an event recorder will be performed at any time if the patient complains of symptoms
Efficacy evaluation: clinical recurrence rate | At 24months after medication
  Defined as atrial fibrillation or atrial tachycardia > 30 sec after medication within 2 year. Based on the 2012 ACC/AHA/HRS guidelines, 24-hour Holter ECG monitoring will be performed at 2 month and every 6 months, and ECG and monitoring with a Holter or an event recorder will be performed at any time if the patient complains of symptoms
Safety evaluation: Major cardiovascular event rate after medication | At 2 months after medication
  Death, Hospitalization, Systemic embolism related atrial fibrillation, Cerebrovascular disease, Stroke, Hemorrhage
Safety evaluation: Major cardiovascular event rate after medication | At 6 months after mediation
  Death, Hospitalization, Systemic embolism related atrial fibrillation, Cerebrovascular disease, Stroke, Hemorrhage
Safety evaluation: Major cardiovascular event rate after medication | At 12 months after mediacation
  Death, Hospitalization, Systemic embolism related atrial fibrillation, Cerebrovascular disease, Stroke, Hemorrhage
Safety evaluation: Major cardiovascular event rate after medication | At 18 months after mediacation
  Death, Hospitalization, Systemic embolism related atrial fibrillation, Cerebrovascular disease, Stroke, Hemorrhage
Safety evaluation: Major cardiovascular event rate after medication | At 24 months after mediacation
  Death, Hospitalization, Systemic embolism related atrial fibrillation, Cerebrovascular disease, Stroke, Hemorrhage

SECONDARY OUTCOMES:
Comparison of cardioversion frequency | At 2 months after medication
  comparison of cardioversion fequency after medication (including re-hospitalization for complication by heart failure, embolism and hemorrhage)
Comparison of cardioversion frequency | At 6 months after medication
  comparison of cardioversion fequency after medication (including re-hospitalization for complication by heart failure, embolism and hemorrhage)
Comparison of cardioversion frequency | At 12 months after medication
  comparison of cardioversion fequency after medication (including re-hospitalization for complication by heart failure, embolism and hemorrhage)
Comparison of cardioversion frequency | At 18 months after medication
  comparison of cardioversion fequency after medication (including re-hospitalization for complication by heart failure, embolism and hemorrhage)
Comparison of cardioversion frequency | At 24 months after medication
  comparison of cardioversion fequency after medication (including re-hospitalization for complication by heart failure, embolism and hemorrhage)
re-ablation(RFCA) fequency | At 2 months after medication
  re-ablation(RFCA) fequency after medication.
re-ablation(RFCA) fequency | At 6 months after medication
  re-ablation(RFCA) fequency after medication.
re-ablation(RFCA) fequency | At 12 months after medication
  re-ablation(RFCA) fequency after medication.
re-ablation(RFCA) fequency | At 18 months after medication
  re-ablation(RFCA) fequency after medication.
re-ablation(RFCA) fequency | At 24months after medication
  re-ablation(RFCA) fequency after medication.
Rate of re-hospitalization | At 2 months after medication
  Rate of re-hospitalization after medication
Rate of re-hospitalization | At 6 months after medication
  Rate of re-hospitalization after medication
Rate of re-hospitalization | At 12 months after medication
  Rate of re-hospitalization after medication
Rate of re-hospitalization | At 18 months after medication
  Rate of re-hospitalization after medication
Rate of re-hospitalization | At 24 months after medication
  Rate of re-hospitalization after medication
Frequency of drug complication | At 2 months after medication
  Frequency of drug complication after medication
Frequency of drug complication | At 6 months after medication
  Frequency of drug complication after medication
Frequency of drug complication | At 12 months after medication
  Frequency of drug complication after medication
Frequency of drug complication | At 18 months after medication
  Frequency of drug complication after medication
Frequency of drug complication | At 24 months after medication
  Frequency of drug complication after medication
Rate of discontinuation of medication | At 2 months after medication
  Rate of discontinuation of medication due to complication
Rate of discontinuation of medication | At 6 months after medication
  Rate of discontinuation of medication due to complication
Rate of discontinuation of medication | At 12 months after medication
  Rate of discontinuation of medication due to complication
Rate of discontinuation of medication | At 18 months after medication
  Rate of discontinuation of medication due to complication
Rate of discontinuation of medication | At 24 months after medication
  Rate of discontinuation of medication due to complication

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided